CLINICAL TRIAL: NCT00554814
Title: Interest of Biofer ® Compound Used in Blédilait Follow on Milk and Growing Milk on Iron Status Evolution in Infant With Latent Iron Deficiency
Brief Title: Interest of Biofer ® Compound Used in Blédilait Follow on Milk in Infant With Latent Iron Deficiency
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: Bledina (Industry)
Responsible Party: Valérie BRENAS, Bledina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BL010; N° ID RCB : 2007-A00684-49
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Last update posted 2008-11-17 (Estimated); Status verified 2008-11

CONDITIONS: Latent Iron Deficiency
Keywords: Iron deficiency; Ferritin; Encapsulated iron; Infant formula
MeSH Terms: conditions — Iron Deficiencies | interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 3 (Experimental): Blédilait Biofer® milk (1,1mg/100kcal)
  Interventions: Drug: Blédilait Biofer®
- 1 (Experimental): Blédilait Biofer® milk (2mg/100kcal)
  Interventions: Drug: Bledilait Biofer®
- 2 (Active Comparator): Milk supplemented with ferrous sulphate (2mg/100kcal)
  Interventions: Drug: Milk supplemented with ferrous sulphate

INTERVENTIONS:
Drug: Bledilait Biofer® — Bledilait Biofer® 2 mg/100 kcal
  Arms: 1
Drug: Milk supplemented with ferrous sulphate — Milk supplemented with ferrous sulphate (2mg/100kcal)
  Arms: 2
Drug: Blédilait Biofer® — Blédilait Biofer® milk (1,1mg/100kcal)
  Arms: 3

SUMMARY:
The primary purpose of the study is to demonstrate the superiority of Bledilait milk (Biofer® 2mg/100kcal) in comparison with ferrous sulphate supplemented milk (2 mg/100 kcal) in infants (6 to 12 months) with latent iron deficiency by measuring serum ferritin value after 2 months of consumption of studied milks.

ELIGIBILITY:
Inclusion Criteria:

* infant between 6 and 12 months of age,
* preterm infant, low birth weight infant (< 2,5 kg), multiple pregnancy, infant from mother with close pregnancies (2 babies in 2 years),
* infant with a serum ferritin value < 12ng/ml and with a normal haemoglobin value (> 11 g/dl), i.e. with a latent iron deficiency,
* infant whose parents or legal tutors have given written informed consent,
* parents or legal tutors agreeing for 4 month follow-up by the investigator,
* infant for which a clinical exam has been performed,
* infant with health insurance.

Exclusion Criteria:

* infant with serum ferritin value < 12 ng/ml and haemoglobin value < 11 g/dl
* infant already receiving medicinal iron supplementation,
* infant with acquired or congenital defect,
* infant presenting a significant metabolic, organic or digestive disease able to interfere with study (including hemochromatosis)
* infant with congenital and/or chromosomal malformation
* infant receiving a drug susceptible, according to the investigator, to interfere with the measured study parameters
* infant needing specific infant formula (hypoallergenic, without cow milk proteins)
* infant in a situation that could, according to investigator, interfere with an optimal participation to the study or be a health risk

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 249 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-11 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Serum ferritin value measured after 2 months of studied milks consumption. | 2 months

SECONDARY OUTCOMES:
- Serum ferritin value - Serum ferritin evolution - CMV evolution - Red blood cells evolution - Common Infectious diseases - Antibiotic consumption | baseline, baseline + 2 months, baseline + 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacques LANGUE, Principal Investigator
Locations (1):
- Alain BOCQUET, Besançon, France

REFERENCES:
- [Derived] Rughwani H, Singh AP, Ramchandani M, Jagtap N, Pal P, Inavolu P, Reddy PM, Januszewicz W, Sekaran A, Nabi Z, Patel R, Lakhtakia S, Banerjee R, Memon SF, Balram P, Darishetty S, Rao GV, Reddy DN. A Randomized, Controlled Trial Comparing the Total Enteroscopy Rate and Diagnostic Efficacy of Novel Motorized Spiral Enteroscopy and Single-Balloon Enteroscopy in Patients With Small-Bowel Disorders: The Motor Trial (NCT 05548140). Am J Gastroenterol. 2023 Oct 1;118(10):1855-1863. doi: 10.14309/ajg.0000000000002409. Epub 2023 Jul 19. PMID 37463435